CLINICAL TRIAL: NCT01153867
Title: Schema-Focused Therapy for Chronic Depression: Efficacy and Mechanisms of Change
Brief Title: Schema Focused Therapy for Chronic Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Academic Community Mental Health Centre (RIAGG) (Other)
Responsible Party: Principal Investigator, Fritz Renner, Dr, Maastricht University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEC 10-3-048
Record Dates: First submitted 2010-06-29; First posted 2010-06-30 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Chronic Major Depressive Disorder
Keywords: Schema Focused Therapy; Chronic Depression; Mechanisms of Change

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Schema Focused Therapy (Experimental): Participants will receive Schema Focused Therapy
  Interventions: Behavioral: Schema Focused Therapy

INTERVENTIONS:
Behavioral: Schema Focused Therapy — SFT is a novel treatment approach to chronic, lifelong problems that incorporates cognitive, behavioral, experiential and psychodynamic elements and techniques. In the present study participants will receive up to 75 individual sessions of SFT depending on the individual progress in therapy.

SUMMARY:
Schema focused therapy (SFT) is an innovative treatment approach to chronic, lifelong problems that incorporates cognitive, behavioral, experiential and psychodynamic elements and techniques. This study will determine whether SFT is a suitable and effective treatment for chronic depression in terms of acute effects and the prevention of relapse/recurrence. The secondary aim of this study is to identify the underlying mechanisms of change in SFT that lead to recovery from depression and the prevention of future relapse/recurrence.

DETAILED DESCRIPTION:
A single-case series design with multiple randomized baselines across participants will be used in this study. The study will last approximately 36 months and comprises three phases. The first phase is a 6-12 weeks waiting list/baseline phase during which participants will be repeatedly assessed with the main outcome measures and putative mediators. In the second phase participants will receive up to 75 individual sessions of SFT for chronic depression depending on the individual progress in therapy. Upon completion of the intervention phase, participants will have monthly follow-up assessments for the next 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Chronic MDD as defined by the DSM-IV (meeting full criteria of MDD for at least 2 years).
* Beck Depression Inventory II (BDI-II) score at screening >=20 (moderate to severe depression)
* Can understand and speak the Dutch language
* Has internet access at home

Exclusion Criteria:

* Acute suicide risk
* Substance induced mood disorder
* Medical condition causes depression directly or through medication intake
* MDD with psychotic features
* DSM-IV Bipolar disorder (current or past)
* DSM-IV Psychotic disorder (current or past)
* DSM-IV alcohol or drug dependence
* Autism Spectrum Disorders (Autistic Disorder, Asperger Syndrome, Pervasive developmental disorder NOS, Rett syndrome, Childhood disintegrative disorder)
* Cluster A and Cluster B personality disorders
* Started with antidepressant medication within three months prior to initial screening. Patients who receive antidepressant medication for more than 3 months prior to the start of the study can keep taking their medication and will not be excluded from participation.
* MRI contra-indications, such as claustrophobia, metal parts in the body and, for women, current pregnancy or breastfeeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Depressive symptom improvement | Weekly during baseline and intervention; Monthly during follow-up

SECONDARY OUTCOMES:
Depressive relapse/recurrence | Measured at 12 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Fritz Renner, PhD, Principal Investigator — Department of Clinical Psychological Science, Maastricht University; Marcus Huibers, PhD, Study Director — Department of Clinical Psychological Science, Maastricht University
Locations (1):
- Academic Community Mental Health Center, Riagg, Maastricht, Limburg, Netherlands